CLINICAL TRIAL: NCT01560767
Title: Can Periarticular Knee Injection of Multimodal Agents Levobupivicaine, Morphine, Ketorolac and Adrenaline Improve Postoperative Pain and Function Following Primary Total Knee Arthroplasty?
Brief Title: Perioperative Analgesia for Knee Arthroplasty (PAKA)
Acronym: PAKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Warwick (Other)
Responsible Party: Principal Investigator, Matthew Costa, Professor of Trauma and Orthopaedic Surgery, University of Warwick
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: PAKA/PROTOCOL/V002; 2010-020466-18 (EudraCT Number)
Record Dates: First submitted 2011-08-16; First posted 2012-03-22 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Knee Arthritis
Keywords: Pain relief; Arthroplasty; periarticular knee infiltration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral Nerve Block (Active Comparator): levobupivacaine
  Interventions: Drug: Femoral Nerve Block
- peri-articular infiltration (Active Comparator): The peri-articular infiltration of multimodal agents will consist of 150 mg of levobupivacaine, 10 mg morphine and 30mg ketorolac diluted in 0.9% saline to make a volume 100 ml. (0.5ml 1:1000 adrenaline will be added to the mixture to reduce blood loss after the operation) Fifty ml of the mixture will be injected into the posterior, medial and lateral soft-tissues just prior to implantation of the TKA components. Care will be taken to avoid excessive infiltration in the area of the common peroneal nerve. Then, while the cement is curing, the anterior soft-tissues including the quadriceps mechanism, the retinacular tissues and the subcuticular tissues will be infiltrated with the remaining 50 ml of peri-articular injection.
  Interventions: Drug: peri-articular infiltration

INTERVENTIONS:
Drug: Femoral Nerve Block — Under aseptic conditions, the femoral artery will be palpated immediately below the inguinal ligament and nerve stimulation will be used to identify the femoral nerve just lateral to the artery. Once the femoral nerve has been identified the block may be performed in the routine manner, using 30 ml of levobupivacaine 0.25%. The precise technique used will be noted on trial documentation.
  Arms: Femoral Nerve Block
Drug: peri-articular infiltration — The peri-articular infiltration of multimodal agents will consist of 150 mg of levobupivacaine, 10 mg morphine and 30mg ketorolac diluted in 0.9% saline to make a volume 100 ml. (0.5ml 1:1000 adrenaline will be added to the mixture to reduce blood loss after the operation) Fifty ml of the mixture will be injected into the posterior, medial and lateral soft-tissues just prior to implantation of the TKA components. Care will be taken to avoid excessive infiltration in the area of the common peroneal nerve. Then, while the cement is curing, the anterior soft-tissues including the quadriceps mechanism, the retinacular tissues and the subcuticular tissues will be infiltrated with the remaining 50 ml of peri-articular injection.
  Arms: peri-articular infiltration

SUMMARY:
Peri-articular knee infiltration with Levobupivicaine 150mg, Morphine 10mg and Ketorolac 30mg reduces postoperative pain following primary total knee replacement compared with the current standard treatment of femoral nerve blockade.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing an elective primary unilateral total knee arthroplasty (TKA) under the care of an orthopaedic consultant at University Hospitals Coventry and Warwickshire NHS trust are potentially eligible for the trial.

Exclusion Criteria:

* Those with sufficient cognitive impairment that they would be unable complete questionnaire (cognitive impairment).
* Those patients who lack capacity under the Mental Capacity Act 2005
* Those patients with a pre-operative history of neurological abnormality in the ipsilateral leg e.g. history of stroke, neurogenic pain or previous nerve injury.
* Those patients having spinal anaesthesia.
* Those patients with a specific contraindication to the analgesic agents used:Morphine: Hypersensitivity reaction Ketorolac: Active or previous peptic ulcer. History of upper gastrointestinal bleeding or perforation, related to previous NSAID therapy.
* Haemorrhagic diatheses, including coagulation disorders
* Hypersensitivity to ketorolac trometamol or other NSAIDs
* Moderate or severe renal impairment (serum creatinine > 160 micromol/l)
* Levobupivicaine: Levobupivacaine solutions are contra-indicated in patients with a known hypersensitivity to levobupivacaine, local anaesthetics of the amide type or any of the excipients
* Uncontrolled angina
* 2nd/ 3rd degree heart block

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 18 Hours post operatively
  A validated, patient-reported 100 mm visual analogue pain score. It is a line 100mm long on which patient places a line through to mark the severity of the pain the patient is experiencing from 0mm= No pain to 100mm wost pain possible.

SECONDARY OUTCOMES:
4 point pain score | First 48 hours post surgery
  An ordinal 4-point pain score recorded every six hours by an independent nurse during the first 48 hrs after the surgery.
Analgesia required | 48 hour period post operativley
  The total use of "as required" analgesia in the first 48hrs after the operation
Concentration of Levobupivicaine in drain and patient serum samples | 6 hours post operation and pre and post retransfusion
  The concentration of local anaesthetic agent (Levobupivicaine) in the drain fluid collected in the Bellovac ABT and patient serum concentrations. The drain concentration will be assessed at 6 hrs post operation with serum concentrations pre-retransfusion (tourniquet- down time + 40 mins) and post-retransfusion (post-op + 6hrs 40min).
Functional Assessments change over time 18, 48 & 6 weeks | 18 & 48 Hours and 6 weeks post surgery
  The patients 'straight-leg raise' and mobilisation will be assessed by an independent physiotherapist on the ward after the surgery and a more formal functional assessment of the knee will be made at 6 weeks using the Oxford Knee Score: a validated, patient-reported measure of knee function.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Costa, Principal Investigator — University of Warwick
Locations (1):
- University of Warwick, University House,, Coventry, United Kingdom